CLINICAL TRIAL: NCT04023409
Title: The Identification of Phenotypes in Patients With Severe Chronic Obstructive Pulmonary Disease (Groningen Severe COPD Cohort)
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Dirk-Jan Slebos, Prof. dr., University Medical Center Groningen
Other Study IDs: NL46286.042.14
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Severe COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe COPD patients: Patients with severe COPD who are referred to the UMCG for a consultation on lung transplantation or bronchoscopic lung volume reduction.
  Interventions: Other: NA: no intervention

INTERVENTIONS:
Other: NA: no intervention — NA: no intervention

SUMMARY:
Rationale: Chronic Obstructive Pulmonary Disease (COPD) is defined by airway obstruction. However, the degree of airflow limitation does not adequately describe the complexity of COPD because significant heterogeneity exists between patients with respect to their clinical presentation, physiology, imaging, response to therapy, decline in lung function and survival. Currently, a clear alternative for describing COPD does not exist but the identification of subgroups of COPD patients based on clinical or genomic and epigenomic factors (phenotypes) could be useful. The continuous flow of very severe COPD patients to the UMCG gives the investigators the unique opportunity to perform a study on the phenotypes of very severe COPD and the underlying gene-environment interaction. The investigators anticipate that the findings of this study will lead to an earlier identification of those subjects who are at risk to develop severe or very severe COPD. In addition, it will lead to a better clinical characterisation of established COPD, possibly enabling a more tailored treatment of different COPD subphenotypes.

Objectives:

Primary Objective:

To identify new clinical phenotypes in patients with severe chronic obstructive pulmonary disease (COPD) using a cluster analysis.

Secondary Objectives:

To:

* identify clinical phenotypes (based on e.g. lung function, clinical, radiologic, systemic, pathological and immunological parameters) in patients with severe COPD.
* identify endotypes/ intermediate phenotypes in patients with severe COPD.
* investigate the contribution of (epi)genomics (including genetics and gene expression) to characterize patients with subsets of severe COPD.

Study design: Observational cross-sectional study with a 2 phase design

Study population: Patients with severe COPD who are referred to the UMCG for a consultation on lung transplantation or bronchoscopic lung volume reduction.

DETAILED DESCRIPTION:
Rationale: Chronic Obstructive Pulmonary Disease (COPD) is defined by airway obstruction. However, the degree of airflow limitation does not adequately describe the complexity of COPD because significant heterogeneity exists between patients with respect to their clinical presentation, physiology, imaging, response to therapy, decline in lung function and survival. Currently, a clear alternative for describing COPD does not exist but the identification of subgroups of COPD patients based on clinical or genomic and epigenomic factors (phenotypes) could be useful. The continuous flow of very severe COPD patients to the UMCG gives the investigators the unique opportunity to perform a study on the phenotypes of very severe COPD and the underlying gene-environment interaction. The investigators anticipate that the findings of this study will lead to an earlier identification of those subjects who are at risk to develop severe or very severe COPD. In addition, it will lead to a better clinical characterisation of established COPD, possibly enabling a more tailored treatment of different COPD subphenotypes.

Objectives:

Primary Objective:

To identify new clinical phenotypes in patients with severe chronic obstructive pulmonary disease (COPD) using a cluster analysis.

Secondary Objectives:

To:

* identify clinical phenotypes (based on e.g. lung function, clinical, radiologic, systemic, pathological and immunological parameters) in patients with severe COPD.
* identify endotypes/ intermediate phenotypes in patients with severe COPD.
* investigate the contribution of (epi)genomics (including genetics and gene expression) to characterize patients with subsets of severe COPD.

Study design: Observational cross-sectional study with a 2 phase design

Study population: Patients with severe COPD who are referred to the UMCG for a consultation on lung transplantation or bronchoscopic lung volume reduction.

Main study parameters: The main study parameter is the identification of new clinical phenotypes. The collected data will allow us to identify new phenotypes, clusters of patients with comparable characteristics. These phenotypes are potentially based on a combination of lung function, clinical, radiologic, systemic and genomic parameters and endotypes, in patients with severe COPD.

ELIGIBILITY:
Inclusion Criteria:

* Referral to the LVR intervention team or LTx team of the (UMCG).
* Chronic Obstructive Pulmonary Disease (COPD) according the Global initiative for Chronic Obstructive Lung Disease (GOLD) criteria (post bronchodilator FEV1/FVC < 0.7)[1]
* Written informed consent.

Exclusion Criteria:

- There are no exclusion criteria for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with severe COPD who are referred to the UMCG for a consultation on lung transplantation or bronchoscopic lung volume reduction.
Sampling Method: Probability Sample
Enrollment: 1030 (Actual)
Dates: Start 2014-08-18 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
clinical phenotypes | baseline
  To identify new clinical phenotypes in patients with severe chronic obstructive pulmonary disease (COPD) using a cluster analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk-Jan Slebos, MD PhD, Principal Investigator — University Medical Center Groningen

IPD SHARING:
Plan to Share IPD: Undecided
Only on request

REFERENCES:
- [Derived] Kuks PJM, Hartman JE, Ter Haar EAMD, van Pelt LJ, Slebos DJ, van den Berge M, Pouwels SD. Identification of Clinically Distinct Clusters in Patients With Severe COPD Using Circulating Blood Cell Population Parameters. Respirology. 2025 Oct 19. doi: 10.1002/resp.70146. Online ahead of print. PMID 41111194
- [Derived] Boersma R, Bakker JT, de Vries M, Raveling T, Slebos DJ, Wijkstra PJ, Hartman JE, Duiverman ML. Defining a phenotype of severe COPD patients who develop chronic hypercapnia. Respir Med. 2024 Nov-Dec;234:107850. doi: 10.1016/j.rmed.2024.107850. Epub 2024 Oct 31. PMID 39488255

DOCUMENTS (1):
  • Study Protocol (2024-06-11): https://cdn.clinicaltrials.gov/large-docs/09/NCT04023409/Prot_000.pdf